CLINICAL TRIAL: NCT04393090
Title: Multiple Myeloma Patients and Their HCPs Tested eHealth Support
Brief Title: eHealth for the Elderly
Acronym: My-eStEPs
Status: Completed | Type: Observational
Sponsor: Cankado GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CAN-17-01
Record Dates: First submitted 2020-05-04; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: eHealth platform CANKADO — The patients were asked to use the open eHealth platform CANKADO as a digital supporting tool.

SUMMARY:
Since internet usage as a complementing element in cancer care is becoming more and more important in oncological routine we launched My-eStEPs (eHealth Strategy for Elderly Patients with Multiple Myeloma) to investigate how specifically elderly patients and their Healthcare Professionals (HCPs) adopt electronic Health (eHealth) support during outpatient treatment. The purpose of this project is to explore how eHealth support influences patients' interaction with their HCPs and how both can benefit from this.

ELIGIBILITY:
Inclusion Criteria:

* multiple myeloma patients
* treated by oral IMiDs

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30 patients (median age 75 years) suffering from multiple myeloma treated by oral IMiDs in 8 medical centers were asked to use the open eHealth platform CANKADO as a digital therapy-supporting tool.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Frequency of patient's internet use | 3 months
  Evaluated in the following criteria: daily, at least once per week, at least once per month, less than once per month
Purpose of patient's internet use | 3 months
  Evaluated in the following criteria: news, online-banking, information collection about products, health-related topics, software downloads, dictionaries
Patient's internet use for health-related topics | 3 months
  Evaluated in the following criteria: does the patient use the internet for health-related topics and if yes, for what exactly
Patient's technical equipment | 3 months
  The presence of following equipment was evaluated: fixed network telephone, smartphone, internet-enabled computer, notebook, laptop, iPad and tablet ownership.
eHealth usage satisfaction | 3 months
  By a structured interview with the patients about their user satisfaction (graded between 1 (best) and 5 (worst))

CONTACTS AND LOCATIONS:
Overall Officials: Timo Schinköthe, PhD, Study Director — Cankado GmbH
Locations (8):
- Germany (8):
  - Hämato-Onkologische Schwerpunktpraxis, Aschaffenburg
  - Onkologie-Köln,, Cologne
  - St.-Antonius-Hospital, Eschweiler
  - Praxis am Albertinen- Krankenhaus, Hamburg
  - Institut für Versorgungsforschung in der Onkologie GbR, Koblenz
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Langen
  - Praxis Dr. med. Peter Ehscheidt, Facharzt für Innere Medizin, Hämatologie, Onkologie, Medikamentöse Tumortherapie und Palliativmedizin, Neuwied
  - Medicum, Wiesbaden